CLINICAL TRIAL: NCT00148200
Title: Prevalence of Female Sexual Dysfunctions Among Healthy Women Coming to the University of Bologna Gynecology Clinic as Outpatients.
Brief Title: Female Sexual Dysfunction: Prevalence Among Italian Healthy Women
Status: Completed | Type: Observational
Sponsor: Unita Complessa di Ostetricia e Ginecologia (Other)
Responsible Party: Dr Maria Cristina Meriggiola, Unita Complessa di Ostetricia e Ginecologia
Other Study IDs: FSD/2005
Record Dates: First submitted 2005-09-02; First posted 2005-09-07 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Sexual Dysfunctions, Psychological
Keywords: female sexual dysfunction; desire; arousal; lubrification; orgasm; satisfaction; pain
MeSH Terms: conditions — Sexual Dysfunctions, Psychological; Orgasm; Personal Satisfaction; Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

SUMMARY:
Purposes of this study are:

* To determine the prevalence of female sexual dysfunctions among Italian general population
* To determine which sexual domains are more frequently compromised
* To evaluate which of the factors we took into consideration are more frequently associated with FSD

DETAILED DESCRIPTION:
BACKGROUND:

Female Sexual Dysfunctions (FSD) are a relatively new field of study as are possible interventions. Until recently FSD were regarded as only a psychological matter and consequently the exact definition of the problem was to some extent controversial. Things have changed and now we refer to FSD according to the classification decided during the International Consensus development Conference on FSD (Basson et al, 2000). There are 5 major categories of FSD: Sexual Desire Disorders, Sexual Arousal Disorders, Orgasmic Disorders, Sexual Pain Disorders. A woman can be considered sexually dysfunctional if she has one or more of these disorders and if she feels uncomfortable about them.

Recent studies completed abroad show the prevalence of FSD to be extremely high: from 38% to 63% of women interviewed about their sexuality have complaints about it.

RATIONALE:

So far, in Italy there are no studies showing the prevalence of FSD among healthy women. We have no reasons to think that the results will demonstrate lower percentages than those found abroad indicating therefore a high number of women complaining about their sexuality.

To define the prevalence of alteration in sexual function we decided to use a questionnaire that would explore all the area included in the definition of FSD. We chose the Female Sexual Function Index (Rosen et al, 2000). This is commonly recognized as a reliable and specific instrument. Moreover there is a validated Italian translation of it.

Women coming to the Gynecologic Clinic for routine examination represent in our opinion a realistic sample of Italian female population.

Complete anonymity will be guaranteed for the entire study to every woman filling out the questionnaire.

During this study we will try to answer the following questions:

* What is the prevalence of FSD among healthy Italian women?
* Which domains of sexuality are most frequently compromised?
* Which among the following factors effect the most sexual functions?
* Age?
* Menopause?
* Stable relationship?
* Duration and quality of relationship?
* Clinical background?
* Reasons for coming to the gynecologic clinic?

DESIGN:

In order to answer these questions the study will be organized as follow

* Request for approval of the study from the local board
* Distribution of the FSFI Questionnaire to female outpatient of the Bologna University Gynecologic Clinic. We are planning to hand ouas many questionnaires as needed to have a minimum of 500 questionnaires completed.
* Registration and analysis of the data from the questionnaires.

MATERIALS AND METHODS:

The FSFI is a multidimensional questionnaire organized into 19 multiple-choice questions and divided in 6 domains which explore sexual desire, arousal, vaginal lubrication, satisfaction and sexual pain. It contains questions about sexual life in the previous 4 weeks. Each answer is given a score between 0 and 5. The final total score gives the result of the test, when it's lower than 26.5 (Wiegel et al, 2005) it suggests a possible sexual dysfunction. FSFI is easily understandable and the time required to complete it is less than 5 minutes.

In our study the FSFI Questionnaire is utilized in conjunction with anonymous questions about age, marital/partner status, duration of relationship, current and past clinical complains, reason for coming to the Gynecologic Clinic and menopause. These will give us the instruments to evaluate whether these factors can influence the presence of FSD and which domains they affect the most.

The questionnaires will be handled by medical staff. The research subjects will be reassured about the anonymity of the study, will be invited to leave the completed FSFI in the collection boxes.

SELECTION OF STUDY POPULATION Selecting women coming for routing testing/exams at the Gynecology Clinic gives us the chance to have our questionnaires completed by a broad sample of women. At least in Italy, where the National Health System guarantees an easy and affordable access to sanitary services, women of all ages and social classes periodically come to clinic to have their gynecologic exam or pap test done. Therefore, even if selected inside a clinic our female sample can reasonably be considered a realistic example of the general female population.

ELIGIBILITY:
Inclusion Criteria:

* Female outpatient coming to Gynecology Clinic
* Age >18

Exclusion Criteria:

* Pregnancy
* Never had sexual activity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: n° 500 Female outpatient coming to Gynecology Clinic
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2005-02; Primary Completion 2006-11 (Actual); Study Completion 2007-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Maria Cristina Meriggiola, MD, Principal Investigator — University of Bologna
Locations (1):
- Clinic of Obstetrics and Gynecology - S. Orsola Hospital, Bologna, Italy

REFERENCES:
- [Background] Laumann EO, Paik A, Rosen RC. Sexual dysfunction in the United States: prevalence and predictors. JAMA. 1999 Feb 10;281(6):537-44. doi: 10.1001/jama.281.6.537. PMID 10022110
- [Background] Basson R, Berman J, Burnett A, Derogatis L, Ferguson D, Fourcroy J, Goldstein I, Graziottin A, Heiman J, Laan E, Leiblum S, Padma-Nathan H, Rosen R, Segraves K, Segraves RT, Shabsigh R, Sipski M, Wagner G, Whipple B. Report of the international consensus development conference on female sexual dysfunction: definitions and classifications. J Urol. 2000 Mar;163(3):888-93. PMID 10688001
- [Background] Berman JR, Berman LA, Werbin TJ, Goldstein I. Female sexual dysfunction: anatomy, physiology, evaluation and treatment options. Curr Opin Urol. 1999 Nov;9(6):563-8. doi: 10.1097/00042307-199911000-00012. PMID 10668578
- [Background] Geiss IM, Umek WH, Dungl A, Sam C, Riss P, Hanzal E. Prevalence of female sexual dysfunction in gynecologic and urogynecologic patients according to the international consensus classification. Urology. 2003 Sep;62(3):514-8. doi: 10.1016/s0090-4295(03)00487-4. PMID 12946757
- [Background] Abdo CH, Oliveira WM Jr, Moreira ED Jr, Fittipaldi JA. Prevalence of sexual dysfunctions and correlated conditions in a sample of Brazilian women--results of the Brazilian study on sexual behavior (BSSB). Int J Impot Res. 2004 Apr;16(2):160-6. doi: 10.1038/sj.ijir.3901198. PMID 14961047
- [Background] Najman JM, Dunne MP, Boyle FM, Cook MD, Purdie DM. Sexual dysfunction in the Australian population. Aust Fam Physician. 2003 Nov;32(11):951-4. PMID 14650796
- [Background] Salonia A, Munarriz RM, Naspro R, Nappi RE, Briganti A, Chionna R, Federghini F, Mirone V, Rigatti P, Goldstein I, Montorsi F. Women's sexual dysfunction: a pathophysiological review. BJU Int. 2004 May;93(8):1156-64. doi: 10.1111/j.1464-410X.2004.04796.x. No abstract available. PMID 15142131
- [Background] Rosen R, Brown C, Heiman J, Leiblum S, Meston C, Shabsigh R, Ferguson D, D'Agostino R Jr. The Female Sexual Function Index (FSFI): a multidimensional self-report instrument for the assessment of female sexual function. J Sex Marital Ther. 2000 Apr-Jun;26(2):191-208. doi: 10.1080/009262300278597. PMID 10782451
- [Background] Wiegel M, Meston C, Rosen R. The female sexual function index (FSFI): cross-validation and development of clinical cutoff scores. J Sex Marital Ther. 2005 Jan-Feb;31(1):1-20. doi: 10.1080/00926230590475206. PMID 15841702
- [Background] Bancroft J, Loftus J, Long JS. Distress about sex: a national survey of women in heterosexual relationships. Arch Sex Behav. 2003 Jun;32(3):193-208. doi: 10.1023/a:1023420431760. PMID 12807292
- [Background] Lightner DJ. Female sexual dysfunction. Mayo Clin Proc. 2002 Jul;77(7):698-702. doi: 10.4065/77.7.698. PMID 12108607